CLINICAL TRIAL: NCT03787212
Title: MiBo ThermoFlo Lid Temperature Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to safety assessment of the study product
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-6281
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MiBo ThermoFlo / Bruder mask (Experimental): Subjects between the ages of 18 to 80 years will be randomly assigned to 1 of 2 treatment sequences in a contralateral fashion.
  Interventions: Device: MiBo ThermoFlo; Device: Bruder Mask
- Bruder Mask / MiBo ThermoFlo (Experimental): Subjects between the ages of 18 to 80 years will be randomly assigned to 1 of 2 treatment sequences in a contralateral fashion.
  Interventions: Device: MiBo ThermoFlo; Device: Bruder Mask

INTERVENTIONS:
Device: MiBo ThermoFlo — Test Device
Device: Bruder Mask — Control Device

SUMMARY:
This study is a prospective, contralateral, single-site, single-visit unmasked evaluation of external and internal eyelid temperature after treatment with the MiBo ThermoFlo.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Between 18 and 80 (inclusive) years of age at the time of screening.
  4. Subjects must possess a functional/usable pair of spectacles and bring them to the visit (only if applicable - to the investigators discretion).

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or breastfeeding.
  2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with participation in the study.
  3. Clinically significant (Grade 3 or 4 on the FDA classification scale) slit lamp findings (e.g. corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection).
  4. Grade 3-4 Percentage of Partial Meibomian Glands on the Pult 5-point grading scale.
  5. Any active Ocular Infection or Inflammation
  6. Any history of eyelid surgery or abnormality
  7. History of Metal Implants in the Eyelids
  8. Any known hypersensitivity or allergic reaction to ultrasound coupling gel.
  9. LASIK Surgery within 2 weeks of the Baseline Visit.
  10. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  11. History of MiBo ThermoFlo or Lipiflow treatment Within the Last 6 months.
  12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, College of Optometry, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 subjects were enrolled into this study prior to its termination. This study was terminated early by the sponsor due to a warning letter from the FDA regarding non-compliance to 21 CFR part 820.
Groups:
- Test/Control: Subjects randomized to this sequence received the MiBo ThermoFlo as Test in their left eye and then received the Bruder Moist Heat Single Eye Compress as Control in their right eye.
- Control/Test: Subjects randomized to this sequence received the Bruder Moist Heat Single Eye Compress as Control in their left eye and then received the MiBo ThermoFlo as Test in their right eye
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study Termination | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study prior to early study termination.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.25 (7.847)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  White | 3
  Asian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Posterior Eyelid Temperature (Palpebral Conjunctiva)
Description: Ocular surface temperature is usually 34.03±0.51ºC in the normal eye. The temperature required to melt obstructive secretions in the Meibomian glands ranges from 32- 35°C but the more severely obstructed glands present in MGD could require a temperature of >40°C, for effective treatment. there is an approximate 5°C difference in temperature between heat applied on the external eyelid surfaces and that reaches the inner surface of the lids, where the meibomian glands are located. This difference was due to both dissipation of heat while passing through the lid tissues and to constant movement of blood through vasculature wicking heat away from the lids. Therefore, achieving the desired temperature of 40°C at the palpebral conjunctiva requires a constant heat of at least 45°C be maintained on the outer lid surface, a temperature which could be both uncomfortable and risk causing thermal injury to the eyelid skin.
Time Frame: 12-minutes post treatment
Population: All subjects that completed all study visits and did not had a protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: Celcius
Units Other Than Participants: eyes
Groups:
- Test: Subjects that recieved the Test treatment during any point in this study
- Control: Subjects that recieved the Control treatment at any point during this study.
Arm/Group | Test | Control
Number analyzed (Participants) | 3 | 2
Number analyzed (eyes) | 3 | 2
Celcius
  Left Eye - Lower Lid: number analyzed (eyes) | 2 | 0
  Left Eye - Lower Lid | 37.835 (0.9829) |
  Left Eye - Upper Lid: number analyzed (eyes) | 2 | 0
  Left Eye - Upper Lid | 36.545 (0.1485) |
  Right Eye - Lower Lid: number analyzed (eyes) | 1 | 2
  Right Eye - Lower Lid | 37.42 (0) | 37.415 (0.5162)
  Right Eye - Upper Lid: number analyzed (eyes) | 1 | 2
  Right Eye - Upper Lid | 35.77 (0) | 37.19 (0.1131)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 1 day per subject, due to early study Termination.
Groups:
- Control: Subjects that recieved the Control treatment at any point during the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
The study was discontinued by the sponsor, due to the manufacturer of the MiBo ThermoFlo receiving a warning letter from the FDA regarding non-compliance to 21 CFR part 820. Subsequently, the primary analyses were not carried.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03787212/Prot_SAP_000.pdf